CLINICAL TRIAL: NCT05466110
Title: sPinal coRd stimulatiOn coMpared With Lumbar InStrumEntation for Low Back Pain After Previous Lumbar Decompression (PROMISE): a Prospective Randomized Controlled Study
Brief Title: Spinal Cord Stimulation Versus Instrumentation for FBSS
Acronym: PROMISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Augsburg (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0221
Record Dates: First submitted 2022-04-25; First posted 2022-07-20 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2022-04

CONDITIONS: Failed Back Surgery Syndrome; SCS; Neuromodulation; Spinal Cord Stimulation; Spinal Fusion; Low Back Pain
MeSH Terms: conditions — Failed Back Surgery Syndrome; Low Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Spinal Cord Stimulation Device (Experimental): The spinal cord stimulators WaveWriter AlphaTM (Boston Scientific) are designed to treat chronic back or leg pain by electrically stimulating the spinal cord. It is a well established worldwide licensed device. Percutaneous lead(-s) are implanted in the epidural space of the thoracic spine during the initial procedure. After discharge a trial phase is initiated and performed according to local preferences and standard of operations (SOPs). Patients are monitored for any complications and pain reduction. If a significant pain reduction (>50 % on the NRS scale for back pain) is achieved, the permanent implantable pulse generator (IPG) is implanted. Otherwise if the therapy remains non-beneficial throughout the trial phase, the leads will be explanted. Patients are allowed to crossover in the fusion group at any point of time.
  Interventions: Device: Spinal Cord Stimulation
- Control - Lumbar Fusion surgery (Active Comparator): The control group needs to represent the standard of care of current practice. Gold standard is lumbar fusion surgery [Resnik 2005]. Surgical instrumentation will be performed according to local preferences and SOPs. Safety and efficacy of these fusion techniques have been repeatedly proven
  Interventions: Procedure: Spinal Fusion Surgery

INTERVENTIONS:
Device: Spinal Cord Stimulation — Epidural application of electrical current to the spinal cord
  Other Names: SCS
  Arms: Spinal Cord Stimulation Device
Procedure: Spinal Fusion Surgery — screw-rod system based spinal instrumentation
  Arms: Control - Lumbar Fusion surgery

SUMMARY:
Low back pain affects people of all ages and has become the leading cause of living with disability worldwide. Patients, suffering from persistent pain after spinal surgery in the absence of any clear spinal pathology are defined of having a "failed back surgery syndrome (FBSS)" and treatment of FBSS remains a great controversy in the spinal community. Apart from conservative treatment, spinal fusion remains as therapeutic option. Furthermore, minimal invasive Neuromodulation techniques might be a promising alternative. Aim of this randomized interventional multi center study is to compare treatment success in FBSS patients with either spinal cord stimulation (SCS) or fusion surgery, 12 months after intervention according to the Oswestry Disability Index (ODI) and other scales and scores. Radiological and health economic outcome also will be analysed for thorough comparison of techniques. Additionally, the safety of the interventions needs to be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Symptomatic degenerative disc disease with LBP as a predominant symptom for at least 6 months following pervious surgery for disc herniation
* ODI score at least 21
* Correctly signed informed consent form

Exclusion Criteria:

* Spinal stenosis resulting in spinal claudication or neurological deficits
* Spinal Instability (> 3 mm Motion on dynamic Lumbar X-rays)
* Major psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability index / ODI | 12 months after intervention
  A patient reported outcome measure to rate pain and disability

SECONDARY OUTCOMES:
Adverse events | 12 months after intervention
  Comparison of complication rates
SF36 | 12 months after intervention
  Score to assess quality of life
EuroQOL 5D | 12 months after intervention
  Score to assess quality of life
hospital length of stay | through study completion, an average of 2 years
  Time measured in days, counting from the first day of hospitalization until the day of discharge of the hospitalization the surgical intervention was performed. If surgery is performed as staged procedure in two separate hospitalizations (SCS) both hospitalizations are counted as described above and days are summed up.
Crossover rates | 12 months after intervention
  Rates of crossover to another therapy arm
Pain medication | 12 months after intervention
  Amount of analgesics taken (drug, dose, mode of application)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Augsburg Department of Neurosurgery, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resnick DK, Choudhri TF, Dailey AT, Groff MW, Khoo L, Matz PG, Mummaneni P, Watters WC 3rd, Wang J, Walters BC, Hadley MN; American Association of Neurological Surgeons/Congress of Neurological Surgeons. Guidelines for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 10: fusion following decompression in patients with stenosis without spondylolisthesis. J Neurosurg Spine. 2005 Jun;2(6):686-91. doi: 10.3171/spi.2005.2.6.0686. PMID 16028738
- [Background] Brox JI, Sorensen R, Friis A, Nygaard O, Indahl A, Keller A, Ingebrigtsen T, Eriksen HR, Holm I, Koller AK, Riise R, Reikeras O. Randomized clinical trial of lumbar instrumented fusion and cognitive intervention and exercises in patients with chronic low back pain and disc degeneration. Spine (Phila Pa 1976). 2003 Sep 1;28(17):1913-21. doi: 10.1097/01.BRS.0000083234.62751.7A. PMID 12973134
- [Background] Fritzell P, Hagg O, Wessberg P, Nordwall A; Swedish Lumbar Spine Study Group. 2001 Volvo Award Winner in Clinical Studies: Lumbar fusion versus nonsurgical treatment for chronic low back pain: a multicenter randomized controlled trial from the Swedish Lumbar Spine Study Group. Spine (Phila Pa 1976). 2001 Dec 1;26(23):2521-32; discussion 2532-4. doi: 10.1097/00007632-200112010-00002. PMID 11725230
- [Background] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Blood E, Hanscom B, Herkowitz H, Cammisa F, Albert T, Boden SD, Hilibrand A, Goldberg H, Berven S, An H; SPORT Investigators. Surgical versus nonsurgical therapy for lumbar spinal stenosis. N Engl J Med. 2008 Feb 21;358(8):794-810. doi: 10.1056/NEJMoa0707136. PMID 18287602
- [Background] Kapural L, Yu C, Doust MW, Gliner BE, Vallejo R, Sitzman BT, Amirdelfan K, Morgan DM, Brown LL, Yearwood TL, Bundschu R, Burton AW, Yang T, Benyamin R, Burgher AH. Novel 10-kHz High-frequency Therapy (HF10 Therapy) Is Superior to Traditional Low-frequency Spinal Cord Stimulation for the Treatment of Chronic Back and Leg Pain: The SENZA-RCT Randomized Controlled Trial. Anesthesiology. 2015 Oct;123(4):851-60. doi: 10.1097/ALN.0000000000000774. PMID 26218762
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Achttien RJ, Powell A, Zoulas K, Staal JB, Rushton A. Prognostic factors for outcome following lumbar spine fusion surgery: a systematic review and narrative synthesis. Eur Spine J. 2022 Mar;31(3):623-668. doi: 10.1007/s00586-021-07018-5. Epub 2021 Oct 27. PMID 34705106
- [Derived] Krauss P, Motov S, Bonk MN, Prescher A, Scorzin J, Hajiabadi MM, Schulte DM, Sommer B, Seiz-Rosenhagen M, Ahmadi R, Maciaczyk J, Lehmberg J, Shiban E. sPinal coRd stimulatiOn coMpared with lumbar InStrumEntation for low back pain after previous lumbar decompression (PROMISE): a prospective multicentre RCT. BMJ Open. 2023 Apr 3;13(4):e067784. doi: 10.1136/bmjopen-2022-067784. PMID 37012023